CLINICAL TRIAL: NCT07236047
Title: Randomized Controlled Trial Comparing Fistulotomy vs LIFT Plus Laser Ablation vs Open LIFT Plus Laser in the Treatment of Trans-sphincteric Perianal Fistula
Brief Title: Comparing Three Surgical Techniques for the Treatment of Transsphincteric Perianal Fistula: (1) Traditional Fistulotomy (Lay Open), (2) Ligation of the Intersphincteric Tract (LIFT) With Adjunctive Endo Fistula Laser Ablation, and (3) Open LIFT Procedure Followed by LASER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0307609
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-04

CONDITIONS: Perianal Fistula
Keywords: LIFT; perianal fistula; LASER
MeSH Terms: interventions — Lifting; Lasers

STUDY DESIGN:
Intervention Model Description: Title:
  Randomized Controlled Trial Comparing Fistulotomy vs LIFT with Laser Ablation vs Open LIFT plus Laser in the Treatment of Transsphincteric Perianal Fistula
  Objective:
  To compare healing rate, recurrence, pain, and functional outcomes among three surgical techniques for transsphincteric fistula.
  Design:
  Single-center, prospective, randomized controlled trial
  Three parallel arms
  90 participants total (30 per group)
  Inclusion Criteria:
  Adults aged 18-65
  Confirmed diagnosis of transsphincteric cryptoglandular perianal fistula
  Primary (first-time) surgery
  Able to provide informed consent
  Exclusion Criteria:
  Crohn's disease or other inflammatory bowel disease
  Suprasphincteric, extrasphincteric, or horseshoe fistulas
  Previous fistula surgery
  Active perianal abscess
  Current immunosuppression
  Pregnant or breastfeeding women
  Primary Outcome:
  Clinical healing (no discharge, closure of opening) at 6 months
  Secondary Outcomes:
  Recurrence at 12 months
  Postoperative
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lay open (Active Comparator): fistula lay open of the tract
  Interventions: Procedure: fistula lay open
- LIFT plus LASER (Active Comparator): ligation of inters-sphincteric tract plus laser for the outer tract
  Interventions: Procedure: LIFT plus LASER
- open LIFT plus LASER (Active Comparator): cutting internal sphincter and ligation of tract plus LASER to outer part
  Interventions: Procedure: open LIFT plus LASER

INTERVENTIONS:
Procedure: fistula lay open — lay open of fistula tract
  Arms: lay open
Procedure: LIFT plus LASER — ligation of inter-sphincteric tract plus LASER of tract
  Arms: LIFT plus LASER
Procedure: open LIFT plus LASER — cutting of internal anal sphincter plus ligation of inter-sphincteric tract plus LASER
  Arms: open LIFT plus LASER

SUMMARY:
>This randomized clinical trial compares three different surgical techniques for the treatment of transsphincteric perianal fistula: (1) traditional fistulotomy (lay open), (2) ligation of the intersphincteric tract (LIFT) with adjunctive endofistula laser ablation, and (3) open LIFT procedure followed by direct laser ablation of the tract under vision. The aim is to determine which approach offers the highest healing rate, lowest recurrence, and best postoperative outcomes with minimal impact on continence.

DETAILED DESCRIPTION:
> Transsphincteric perianal fistula presents a surgical challenge due to the need to balance fistula eradication with continence preservation. While fistulotomy is associated with high healing rates, it carries a risk of sphincter damage. Ligation of the intersphincteric tract (LIFT) offers a sphincter-sparing alternative, and the use of endofistula laser ablation (FiLaC or diode laser) has shown promise in enhancing outcomes.

This study will enroll 90 patients with confirmed transsphincteric cryptoglandular perianal fistula and randomize them equally into three arms:

Group A: Conventional fistulotomy (lay open).

Group B: LIFT procedure with endofistula laser ablation using a radial laser fiber.

Group C: Open LIFT with direct laser ablation of the tract under vision.

The primary endpoint is complete clinical healing at 6 months. Secondary outcomes include recurrence rates at 12 months, pain scores (VAS), continence outcomes (Wexner score), return to daily activities, and patient satisfaction. The study aims to determine the optimal balance between healing efficacy and preservation of continence.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65
* Confirmed diagnosis of transsphincteric cryptoglandular perianal fistula
* Primary (first-time) surgery
* Able to provide informed consent

Exclusion Criteria:

* Crohn's disease or other inflammatory bowel disease
* Suprasphincteric, extrasphincteric, or horseshoe fistulas
* Previous fistula surgery
* Active perianal abscess
* Current immunosuppression
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
healing | 6 months
  Baseline Fistula manegment score → Pre-op disease severity Post-op Fm-score at 1, 3, 6 months → Objective clinical healing Where Total score = Pain + Discharge + Continence + QOL with Range = 0-16 Pain (0-4) 0 No pain
  1. Mild, occasional pain, no analgesics needed
  2. Moderate pain occasional analgesics
  3. Severe pain regular analgesics
  4. Constant, severe pain interfering with daily activities Discharge (0-4)
  0 No discharge
  1 Occasional spotting, no pad required 2 Daily discharge, small amount, 1 pad/day 3 Moderate discharge requiring >1 pad/day 4 Persistent heavy discharge; soaking pads; malodorous Continence (0-4) 0 Full continence
  1 Gas incontinence only 2 Occasional soiling or minor liquid incontinence 3 Frequent soiling; liquid stool incontinence 4 Solid stool incontinence Quality of Life (QoL) 0 No impact on life
  1. Mild limitation
  2. Moderate impact
  3. Significant impact
  4. Severe impairment Interpretation of healing 0-3 Minimal 4-7 Mild disease
  8 - 11 moderate 12 - 17 severe

SECONDARY OUTCOMES:
Fistula manegment score above 7 consider non healing | 12 months
  Baseline Fistula manegment score → Pre-op disease severity Post-op Fm-score at 12 months → Objective clinical non healing Where Total score = Pain + Discharge + Continence + QOL with Range = 0-16 Pain (0-4) 0 No pain
  1. Mild, occasional pain, no analgesics needed
  2. Moderate pain occasional analgesics
  3. Severe pain regular analgesics
  4. Constant, severe pain interfering with daily activities Discharge (0-4)
  0 No discharge
  1 Occasional spotting, no pad required 2 Daily discharge, small amount, 1 pad/day 3 Moderate discharge requiring >1 pad/day 4 Persistent heavy discharge; soaking pads; malodorous Continence (0-4) 0 Full continence
  1 Gas incontinence only 2 Occasional soiling 3 Frequent soiling 4 Solid stool incontinence Quality of Life (QoL) 0 No impact on life
  1. Mild limitation
  2. Moderate impact
  3. Significant impact
  4. Severe impairment Interpretation of healing 0-3 Minimal 4-7 Mild disease
  8 - 11 moderate 12 - 17 severe Score above 7 consider non healing
continence level. Assessed by wexener incontinence score | 6 months
  Wexner score is clinical tool used to quantify the severity of fecal incontinence. five specific components, and each component is scored from 0 to 4. The total score ranges from 0 to 20, where 0 represents perfect continence and 20 represents complete incontinence.
  Incontinence to solid stool:
  0 means this never occurs.
  1. means it happens rarely (> once a month).
  2. indicates it occurs sometimes (> once a week).
  3. means it happens usually (< once a week).
  4. reflects constant or daily incontinence.
  Incontinence to liquid stool:
  Scored in the same way as solids, from 0 (never) to 4 (always).
  Incontinence to gas:
  scored from 0 to 4 using the same frequency scale.
  Use of pads for protection:
  Scored from 0 (no need for pads) to 4 (pads required all the time). 5. Lifestyle alteration due to incontinence: 0 means no effect on lifesty and 4 sever effect 0: Perfect continence 1-5: Mild incontinence 6-10: Moderate 11-20 severe

CONTACTS AND LOCATIONS:
Overall Officials: Walid GALAL Elshazly, Prof, Principal Investigator — University of Alexandria

IPD SHARING:
Plan to Share IPD: No